CLINICAL TRIAL: NCT01918332
Title: A Multicenter, Randomized, Factorial, Double-blinded, Double-dummy Phase Ⅲ Trial to Evaluate the Efficacy and Safety of the Coadministration of Valsartan 160mg and Rosuvastatin 20mg in Comparison to Each Component Administered Alone in Patients With Hypertension and Hyperlipidemia
Brief Title: Efficacy and Safety of Valsartan 160mg and Rosuvastatin 20mg in Patients With Hypertension and Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: LG-VRCL002
Record Dates: First submitted 2013-08-05; First posted 2013-08-07 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension,; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Valsartan; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Valsartan 160mg, Rosuvastatin 20mg (Experimental): Both Valsartan 160mg and Rosuvastatin 20mg are administered daily by mouth once a day for 8 weeks.
  Interventions: Drug: Valsartan 160mg; Drug: Rosuvastatin 20mg
- Valsartan 160mg, Rosuvastatin 20mg placebo (Active Comparator): Intervention : Drug : Both Valsartan 160mg and Rosuvastatin 20mg placebo are administered daily by p.o. once a day for 8 weeks.
  Interventions: Drug: Valsartan 160mg; Drug: Rosuvastatin 20mg placebo
- Valsartan 160mg placebo, Rosuvastatin 20mg (Active Comparator): Intervention : Drug : Both Valsartan 160mg placebo and Rosuvastatin 20mg are administered daily by p.o. once a day for 8 weeks.
  Interventions: Drug: Rosuvastatin 20mg; Drug: Valsartan 160mg placebo
- Placebo (Placebo Comparator): Intervention : Drug : Both Valsartan 160mg placebo and Rosuvastatin 20mg placebo are administered daily by p.o. once a day for 8 weeks.
  Interventions: Drug: Valsartan 160mg placebo; Drug: Rosuvastatin 20mg placebo

INTERVENTIONS:
Drug: Valsartan 160mg
  Other Names: Diovan
  Arms: Valsartan 160mg, Rosuvastatin 20mg; Valsartan 160mg, Rosuvastatin 20mg placebo
Drug: Rosuvastatin 20mg
  Other Names: Crestor
  Arms: Valsartan 160mg placebo, Rosuvastatin 20mg; Valsartan 160mg, Rosuvastatin 20mg
Drug: Valsartan 160mg placebo
  Arms: Placebo; Valsartan 160mg placebo, Rosuvastatin 20mg
Drug: Rosuvastatin 20mg placebo
  Arms: Placebo; Valsartan 160mg, Rosuvastatin 20mg placebo

SUMMARY:
This study aims to evaluate the efficacy and safety of the coadministration of valsartan (Diovan®) 160mg and rosuvastatin (Crestor®) 20mg in comparison to each component administered alone in patients with hypertension and hyperlipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 20-80 years who has hypertension and hyperlipidemia
2. Patient who has a Hypertension
3. Patient who has a Hyperlipidemia according to NCEP-ATP III guideline(2004)
4. Patient who signed the Informed Consent Form after receiving an explanation on the purpose, methods, and effect of the study

Exclusion Criteria:

1. If blood pressure and fasting serum lipid level measured at screening and Visit 2 (0 week) satisfy the following criteria 1) sitSBP≥180mmHg or sitDBP≥110mmHg (For high risk group, sitSBP≥ 160mmHg or sitDBP ≥100mmHg ) 2) LDL-C>250mg/dL , or TG≥ 400mg/dL
2. If sitSBP difference between the right and left arms >20mmHg or sitDBP difference between the right and left arms > 10mmHg at screening
3. When blood pressure is repeatedly measured from the selected arm at screening, if sitSBP difference ≥ 20mmHg or sitDBP difference ≥10mmHg
4. Patient with orthostatic hypotension accompanying symptoms at screening (decrease in sitDBP ≥10mmHg or decrease in sitSBP ≥ 20mmHg )

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System Severance Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Valsartan 160mg, Rosuvastatin 20mg: Both Valsartan 160mg and Rosuvastatin 20mg are administered daily by mouth once a day for 8 weeks.
  Valsartan 160mg
  Rosuvastatin 20mg
- Valsartan 160mg, Rosuvastatin 20mg Placebo: Intervention : Drug : Both Valsartan 160mg and Rosuvastatin 20mg placebo are administered daily by p.o. once a day for 8 weeks.
  Valsartan 160mg
  Rosuvastatin 20mg placebo
- Valsartan 160mg Placebo, Rosuvastatin 20mg: Intervention : Drug : Both Valsartan 160mg placebo and Rosuvastatin 20mg are administered daily by p.o. once a day for 8 weeks.
  Rosuvastatin 20mg
  Valsartan 160mg placebo
- Placebo: Intervention : Drug : Both Valsartan 160mg placebo and Rosuvastatin 20mg placebo are administered daily by p.o. once a day for 8 weeks.
  Valsartan 160mg placebo
  Rosuvastatin 20mg placebo
Period: Overall Study
Arm/Group | Valsartan 160mg, Rosuvastatin 20mg | Valsartan 160mg, Rosuvastatin 20mg Placebo | Valsartan 160mg Placebo, Rosuvastatin 20mg | Placebo
Started | 43 | 41 | 39 | 45
Completed | 35 | 36 | 30 | 38
Not Completed | 8 | 5 | 9 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3 | 2 | 3
Not completed — Protocol Violation | 6 | 2 | 6 | 3
Not completed — lipid result by central lab did not meet | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan 160mg, Rosuvastatin 20mg | Valsartan 160mg, Rosuvastatin 20mg Placebo | Valsartan 160mg Placebo, Rosuvastatin 20mg | Placebo | Total
Number analyzed (Participants) | 41 | 40 | 35 | 44 | 160
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 21 | 29 | 100
  >=65 years | 15 | 16 | 14 | 15 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 7 | 10 | 47
  Male | 25 | 26 | 28 | 34 | 113

OUTCOME MEASURES:

1. Primary Outcome: sitDBP Changes at Week 8 From Baseline
Description: sitDBP changes of the valsartan 160mg and valsartan placebo groups at Week 8 from baseline
Time Frame: 8 weeks
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- V160+R20 & V160: Valsartan 160mg + Rosuvastatin 20mg & Valsartan 160mg + Rosuvastatin 20mg placebo
- R20 & Placebo: Valsartan 160mg placebo + Rosuvastatin 20mg & Placebo
Arm/Group | V160+R20 & V160 | R20 & Placebo
Number analyzed (Participants) | 81 | 79
mmHg | -9.24 [-10.88 to -7.61] | -2.9 [-4.55 to -1.24]

2. Primary Outcome: LDL-C Percentage Changes at Week 8 From Baseline
Description: LDL-C percentage changes of the rosuvastatin 20mg and rosuvastatin placebo groups at Week 8 from baseline
Time Frame: 8 weeks
Population: FAS
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- V160+R20 & R20: Valsartan 160mg + Rosuvastatin 20mg & Valsartan 160mg placebo + Rosuvastatin 20mg
- V160 & Placebo: Valsartan 160mg + Rosuvastatin 20mg placebo & Placebo
Arm/Group | V160+R20 & R20 | V160 & Placebo
Number analyzed (Participants) | 76 | 84
percent change | -49.91 [-53.34 to -46.47] | -2.38 [-5.65 to 0.88]

ADVERSE EVENTS:
Time Frame: 12~14 weeks (4-6 weeks of Therapeutic Lifestyle Change + 8 weeks of Treatment period)
Description: All adverse events were collected at every visit by interview, physical assessment and laboratory tests .
  The following other AE table presents the subject numbers of AE in the first line in the table and the case numbers of AE in the other rows respectively.
Arm/Group | Valsartan 160mg, Rosuvastatin 20mg | Valsartan 160mg, Rosuvastatin 20mg Placebo | Valsartan 160mg Placebo, Rosuvastatin 20mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/41 | 0/37 | 0/45
Other Adverse Events (participants affected / at risk) | 10/43 | 7/41 | 4/37 | 5/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 160mg, Rosuvastatin 20mg (N=43) | Valsartan 160mg, Rosuvastatin 20mg Placebo (N=41) | Valsartan 160mg Placebo, Rosuvastatin 20mg (N=37) | Placebo (N=45)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 — The subject participated in the study on 17 Sep 2012, and she was randomized on 18 Oct 2012. On that day, the subject had nausea and chest pain after eating cake, and visited the institution and was hospitalized on 22 Oct 2012.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan 160mg, Rosuvastatin 20mg (N=43) | Valsartan 160mg, Rosuvastatin 20mg Placebo (N=41) | Valsartan 160mg Placebo, Rosuvastatin 20mg (N=37) | Placebo (N=45)
conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
nasopharyngisit (Infections and infestations) | 0 | 0 | 0 | 1
nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
asthenia (General disorders) | 0 | 1 | 1 | 0
chest discomfort (General disorders) | 0 | 2 | 0 | 0
chest pain (General disorders) | 0 | 0 | 1 | 0
face oedema (General disorders) | 1 | 0 | 0 | 0
oedema peripheral (General disorders) | 1 | 0 | 0 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 1
aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
blood potassium increased (Investigations) | 0 | 1 | 0 | 0
gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
dizziness (Nervous system disorders) | 1 | 2 | 0 | 0
headache (Nervous system disorders) | 2 | 0 | 0 | 3
hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Withdrawal(discontinuation) leading to smaller number of per-protocol set than full analysis set. The violation of protocol was the criterion of subjects' withdrawal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other